CLINICAL TRIAL: NCT00283972
Title: Health Outcome Study of LAP-BAND Adjustable Gastric Banding System
Brief Title: LAP-BAND Observational Cohort
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Inamed (Industry)
Collaborators: Massachusetts Veterans Epidemiology Research and Information Center (U.S. Federal Agency)
Other Study IDs: 12242004P
Record Dates: First submitted 2006-01-24; First posted 2006-01-31 (Estimated); Last update posted 2006-01-31 (Estimated); Status verified 2006-01

CONDITIONS: Epworth Sleepiness Scale; Glycemic Control; Liver Function; Inflammation; Iron and Bone Turnover; SF-36; IW-QOL Lite HRQoL
Keywords: Health Outcome Study
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: LAP-BAND System

SUMMARY:
To prospectively observe the association of the LAP-BAND procedure on quality of life, anthropometric, metabolic and biochemical parameters in morbidly obese patients when performed by experienced US surgeons. The study will also include a complete economic analysis of the LAP-BAND procedure and follow-up costs Hypothesis: Measurements defining quality of life and the severity of obesity and obesity related comorbidities improve significantly over baseline with the LAP-BAND System treatment at 6 and 12 months post surgery when performed by an experienced surgeon.

DETAILED DESCRIPTION:
Study Type: Observational cohort. Single arm (non-comparative), non-randomized, multi-site surgical case series.

Objective: To prospectively observe the association of the LAP-BAND System device on measurements of quality of life, anthropometric, metabolic and biochemical parameters in morbidly obese patients when performed by experienced U.S. surgeons. Cost effectiveness analysis will also be done.

Numbers: This study will enroll 240 patients total from six U.S. bariatric surgical practices

Duration: Individual subject participation will be approximately 15 months. Data will be collected at a baseline less than three months prior to surgery or before starting a Very Low Calorie Diet (VLCD), then at 6 and 12 months post surgery. The total duration, including enrollment, of the observational period for the cohort is expected to be 21 months. Subjects have the option to consent for future contact by investigators for a period of 10 years following their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Morbid Obesity: BMI >40 kg/m2 or
* BMI > or equal to 35 kg/m2 with significant obesity related comorbidity
* Age 18 years old or older
* Dietary attempts at weight control have been ineffective
* Consented for surgery with LAP-BAND System by pre qualified bariatric surgeon
* Willingness and ability to follow protocol requirements
* Residing within a reasonable distance from the surgeon's office and being able to travel to the surgeon's office to complete all routine follow-up visits

Exclusion Criteria:

* Previous bariatric surgery
* Psychological impairments that would impede compliance with study follow up schedule, as determined by attending surgeons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-06; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Deykin, MD, Study Chair — Massachusetts Veterans Epidemiology Research adn Information Center; Louis Fiore, MD, Principal Investigator — Massachusetts Veterans Epidemiology Research and Information Center